CLINICAL TRIAL: NCT03539198
Title: A Prospective Observational Study of Proton Stereotactic Body Radiation Therapy and Immunotherapy for Recurrent/Progressive Locoregional or Metastatic Head and Neck Cancer
Brief Title: Study of Proton SBRT and Immunotherapy for Recurrent/Progressive Locoregional or Metastatic Head and Neck Cancer
Status: Terminated | Type: Observational
Why Stopped: Failure to accrue.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-010910; ROR1771 (Other: Mayo Clinic)
Record Dates: First submitted 2018-04-30; First posted 2018-05-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiosurgery; Nivolumab; Protons

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Locoregional: Patients with recurrent locoregional head and neck cancer
  Interventions: Radiation: Proton Stereotactic Body Radiation Therapy (SBRT) (5 fractions; 3500-4500 cGy); Drug: Nivolumab 3 mg/kg IV q2 weeks; Radiation: Proton or Photon SBRT (3-5 fractions; various dose and fractionation regimens depending on treatment site).
- Metastatic: Patients with recurrent metastatic head and neck cancer
  Interventions: Radiation: Proton Stereotactic Body Radiation Therapy (SBRT) (3-5 fractions; various dose and fractionation regimens depending on treatment site).; Drug: Nivolumab 3 mg/kg IV q2 weeks; Radiation: Proton or Photon SBRT (3-5 fractions; various dose and fractionation regimens depending on treatment site).

INTERVENTIONS:
Radiation: Proton Stereotactic Body Radiation Therapy (SBRT) (5 fractions; 3500-4500 cGy) — Patients will be receiving proton SBRT
  Groups: Locoregional
Radiation: Proton Stereotactic Body Radiation Therapy (SBRT) (3-5 fractions; various dose and fractionation regimens depending on treatment site). — Patients will receive proton SBRT.
  Groups: Metastatic
Drug: Nivolumab 3 mg/kg IV q2 weeks — Patients will receive Nivolumab x2 cycles before SBRT q2 weeks, and continued q2 weeks after SBRT until progression or at the discretion of the treating physician.
Radiation: Proton or Photon SBRT (3-5 fractions; various dose and fractionation regimens depending on treatment site). — Patients with further oligoprogression (5 or fewer sites) will be eligible to receive additional SBRT to all sites of oligoprogression.

SUMMARY:
This study observes the clinical efficacy of combining proton SBRT with PD-1 blockade immunotherapy in both the locoregionally recurrent and metastatic settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old whose multidisciplinary care team has determined that the treatments outlined in the protocol are the treating physicians' equipoised clinical recommendation, the multidisciplinary head & neck tumor board's recommendation, and that any reasonable alternative treatments have been reviewed with the subject.
* Signed written informed consent in accordance with regulatory and institutional guidelines.
* Must be willing to comply with scheduled visits, treatment schedule, laboratory testing and other study obligations. Patients must be receiving SOC treatment for recurrent or progressive Head and Neck cancer. Please refer to UCM procedural manual.
* Histologically confirmed head and neck squamous cell carcinoma from any of the primary sites: oral cavity, pharynx, larynx, nasopharynx, sinonasal, cutaneous, or unknown head and neck primary.
* Subjects with head and neck squamous cell carcinoma that has progressed during chemotherapy with a platinum-based drug or that has recurred or metastasized after platinum-based chemotherapy or in patients with an intolerance to or contraindication for platinum-based chemotherapy will be eligible.
* ECOG performance status 0-2
* Subjects enrolled on the METASTATIC ARM must have at least two (≥) lesions:

One lesion must be safely amenable to irradiation with stereotactic body radiation therapy per the treating radiation oncologist. Prior radiation to this lesion is allowed if given ≥ 6 months prior. One lesion must be measurable by CT or MRI per iRECIST 1.1 criteria and should be separate from the lesion to be irradiated. If this target lesion has been previously irradiated, there must be documented disease progression after radiation per RECIST 1.1.

* Any prior radiotherapy must have been completed at least 3 weeks prior to enrollment.
* Adequate bone marrow, hepatic, and renal function based on screening lab values within 35 days prior to beginning immunotherapy:

  * WBC ≥ 2 K/microliter
  * Neutrophils ≥ 1.5 K/microliter
  * Platelets ≥ 100 K/microliter
  * Hemoglobin ≥ 9.0 g/deciliter
  * Serum Creatinine ≤ 1.5 x ULN or creatinine clearance > 40ml/min using the Cockcroft-Gault formula.
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
  * AST/ALT ≤ 3 x ULN
  * Total bilirubin <1.5 x ULN (except subjects with Gilbert Syndrome who can have total bilirubin <3.0 mg/deciliter).
* Women of childbearing potential must have a negative serum or urine pregnancy test within 10 days prior to beginning immunotherapy.
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception from time of enrollment for the duration of treatment with nivolumab and for 6 months after discontinuation of nivolumab. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 6 months after the last dose of nivolumab.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Insurance approval or personal pay for SBRT.
* Patient may undergo palliative surgery prior to postoperative proton SBRT and remain in the metastatic arm of the study, as long as the patient meets the other aforementioned criteria relating to the metastatic arm. Surgery is allowable for the locoregionally recurrent arm as per the study schema.

Exclusion Criteria:

* Active brain metastases or leptomeningeal disease. Note: Treated brain metastases (e.g. GammaKnife or surgical resection) are eligible if these have been treated and are without MRI evidence of progression for at least 8 weeks after treatment. MRI must be performed within 35 days prior tobeginning immunotherapy.
* Histologically confirmed non-squamous histologies including salivary gland or other non-squamous histologies (e.g. mucosal melanoma) are not allowed; exception WHO Type I-III nasopharynx, which are allowed.
* Subjects with active autoimmune disease or on steroid therapy of >10 mg/day prednisone or equivalent.
* Subjects who have undergone bone marrow or solid organ transplantation.
* Known HIV, hepatitis B or C infection.
* Treatment with chemotherapy, radiation therapy or immunotherapy including investigational agents within 25 days of beginning immunotherapy.
* Women that are breastfeeding or pregnant.
* Any concurrent chemotherapy, hormonal therapy, immunotherapy, or investigational therapy apart from the prescribed treatment per protocol.
* Other active non-head and neck malignancy <1 year prior to registration. If there is a history of prior distinct malignancy, they must not be receiving chemotherapy, radiotherapy, or immunotherapy for their other disease at the time of protocol enrollment. Exceptions include: Non-melanotic skin cancer and carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with locoregional or metastatic head and neck cancers
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) using iRECIST 1.1 criteria for locoregional arm | From start date of immunotherapy to disease progression; up to 2 years
  ORR is defined as the proportion of patients who achieved a best response of complete response (CR) or partial response (PR) using iRECIST 1.1 criteria, and will be evaluated for both the lesion(s) treated with SBRT, referred to as "Target lesion (+SBRT+Nivo), as well as the lesion(s) not treated with SBRT (if applicable), referred to as "Target lesion (+Nivo only)", per the prescribed treatment. The primary endpoint for the locoregional arm will be considered met if the assumption and desired outcome are achieved for ORR in the "Target lesion(s) (+SBRT+Nivo)". Best overall response (BOR) is defined as the best response designation, recorded between the start date of immunotherapy and the date of progression using iRECIST 1.1 criteria.
Objective response rate (ORR) using iRECIST 1.1 criteria for metastatic arm | From start date of immunotherapy to disease progression; up to 2 years
  ORR is defined as the proportion of patients who achieved a best response of complete response (CR) or partial response (PR) using iRECIST 1.1 criteria, and will be evaluated for both the lesion(s) treated with SBRT, referred to as "Target lesion (+SBRT+Nivo), as well as the lesion(s) not treated with SBRT, referred to as "Target lesion (+Nivo only)", per the prescribed treatment. The primary endpoint for the metastatic arm will be considered met if the assumption and desired outcome are achieved for ORR in the "Target lesion(s) (+Nivo only)" since these are the lesions we hypothesize will have an augmented response from proton SBRT through the abscopal effect. Best overall response (BOR) is defined as the best response designation, recorded between the start date of immunotherapy and the date of progression using iRECIST 1.1 criteria.

SECONDARY OUTCOMES:
Local control rate for both arms | From start date of immunotherapy to disease local progression; up to 1 year
Overall Survival Time for both arms | From start date of immunotherapy to date of death, up to 2 years
Overall Survival for both arms | From start date of immunotherapy to 3, 6, 9, and 12 month
Progression-free survival for both arms | From start date of immunotherapy to disease progression or death, whichever occurs first; assessed up to 2 years
Time to progression (TTP) | From start date of immunotherapy to disease progression, but does not count patients who die from other causes; assessed up to 2 years
New development of distant metastasis for both arms | From start date of immunotherapy to disease progression or death, whichever occurs first; assessed up to 2 years
Quality of Life for both arms | From start date of immunotherapy (baseline evaluation) to approximately 6 months after enrollment at Day 45, 90, 130, and 170
  Quality of life will be assessed through questionaire EORTC QLQ-H&N35
Quality of Life for both arms | From start date of immunotherapy (baseline evaluation) to approximately 6 months after enrollment at Day 45, 90, 130, and 170
  Quality of life will be assessed through questionaire Mayo PRO for Head and Neck
Adverse Effects for both arms | From start date of immunotherapy (baseline evaluation) to approximately 6 months after enrollment at Day 45, 90, 130 and 170
Predictive and prognostic biomarkers for both arms | Baseline, Day 15-30, 45, 90 and 130
  a maximum of 5 blood draws will be used

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Ma, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials